CLINICAL TRIAL: NCT06377475
Title: Herstellung Und Eingliederung Von Michigan-Schienen Durch Zahnmedizinstudierende: Eine Qualitative Und Quantitative Studie
Brief Title: Fabrication and Insertion of Michigan Splints by Dental Students
Status: Enrolling by invitation | Type: Observational
Sponsor: Juliana Marotti Großhausen (Other)
Responsible Party: Sponsor-Investigator, Juliana Marotti Großhausen, PD Dr. med. dent., University of Basel
Organization: University of Basel (Other)
Other Study IDs: 2024-00148; 2024-00148 (Registry Identifier: EKNZ)
Record Dates: First submitted 2024-03-18; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Impression Technic, Dental; Jaw Relationship; Bruxism
Keywords: Bruxism; Jaw Relationship; Impression Technic
MeSH Terms: conditions — Bruxism | interventions — Jaw Relation Record; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wax registration: The jaw relation for the Michigan-splint will be performed with wax.
  Interventions: Procedure: Jaw relation; Procedure: Questionnaire
- JIG registration: The jaw relation for the Michigan-splint will be performed with JIG.
  Interventions: Procedure: Jaw relation; Procedure: Questionnaire

INTERVENTIONS:
Procedure: Jaw relation — The quality of the Michigan-splint will be analyzed according to different interventions (wax or jig jaw relation) and a questionnaire that quantify the occlusal contacts of the splint.
Procedure: Questionnaire — The quality of the Michigan-splint will be analyzed according to different interventions (wax or jig jaw relation) and a questionnaire that quantify the occlusal contacts of the splint.

SUMMARY:
The aim of this study is to investigate the potential effects of different jaw relation determination (KRB) techniques on the fabrication of Michigan splints, in particular by comparing conventional methods with a wax plate and the use of an anterior jig. All materials and methods for the fabrication of the Michigan splint are already part of the curriculum of the Clinic for Dental Prosthodontics for first-year Master-students. Therefore, we intend to conduct a retrospective study (for the 2023 cohort) and a prospective analysis of the data (for the 2024 and 2025 cohorts). Questionnaires, models and intraoral scans will be used to evaluate the efficacy and precision of the different KRB methods as well as the fabrication process of the Michigan splint.

DETAILED DESCRIPTION:
Since its development in the 1960s as a modification of the Sved-biteplane constructed in Scandinavia, the Michigan splint has gained worldwide recognition and can now be described as the gold standard of treatment with stabilization splints for myoarthopathies. The use of stabilization splints - as confirmed in an S3 guideline published by the Association of the Scientific Medical Societies in Germany (AWMF) in 2019 - is classified as a recommendable and, if necessary, reversible therapeutic measure for the treatment of bruxism. As part of a systematic review, additional causes were identified in addition to the seven already known central risk factors for bruxism. In addition to factors such as emotional stress and anxiety disorders, further psychological disorders were added as part of the literature review. Against this background of a predominantly psychologically determined aetiopathogenesis, acceptance of the splint by the patient could represent an important component of successful treatment for bruxism, for example in terms of increased patient compliance. Sufficient evidence-based studies that specifically investigate a possible connection between the type of fabrication of the Michigan splint and its acceptance by the patient are still lacking. The Michigan splint is a proven method for the treatment of patients diagnosed with bruxism. In the conventional method, the KRB of the Michigan splint is fabricated using the wax technique, which can lead to inaccuracies in registration due to its material properties. With the advancement of digital technology, the use of intraoral scanners is becoming more common in dental practices. In these cases, KRB can be performed with a jig using a material with higher precision than wax. Furthermore, the KRB can be scanned with the JIG without interfering with wax. To date, no studies have been conducted comparing the quality of the Michigan splint with these two KRB methods. For the fabrication of the jig, the condyles must serve as support points, which is why it is not possible to perform in vitro studies with the JIG.

The primary objective of this study is to descriptively analyze the quality of Michigan splints fabricated by dental students. The parameters examined relate to the fit, extension and function of the splint. Likewise, the common KRB methods (wax plate and anterior jig) are to be compared in order to identify any discrepancies and thus consequences in the fabrication of the splint. The data obtained from the scans will be analyzed and points compared in order to compare possible differences between the various bite registration methods. The secondary aim of this study is to analyze and possibly improve the fabrication process of Michigan splints in the context of dental student education.

ELIGIBILITY:
Inclusion Criteria:

* Dental students in the first year of their Master's degree
* 18 years and older, gender independent
* Ability to give informed consent, documented by signature

Exclusion Criteria:

* Inability or contraindications (e.g. dental pain, dental mobility, generalized periodontitis, removable denture wearers, acute infection) to undergo the procedure under study
* Inability to follow the procedures of the study, e.g. due to language problems, depression or mental disorders
* Students who do not consent to the analysis of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders are eligible to participate in the study.
Study Population: Dental Students
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Wax vs JIG Registration | From enrollment to the end of treatment at 6 weeks
  The deviation (in micrometers) between the wax and JIG registration will be measured with the software CloudCompare.

SECONDARY OUTCOMES:
Questionnaire | From enrollment to the end of treatment at 6 weeks
  In order to analyze the quality of the splints, a questionnaire will be implemented where points will be given (For example: 0=unsatisfactory, 1=corrections needed, 2=satisfactory) for the each topic and answer.

CONTACTS AND LOCATIONS:
Locations (1):
- UZB, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
I will share the IPD upon request. All data, study protocol and informed consent of participants can be shared.